CLINICAL TRIAL: NCT07260422
Title: EVALUATION OF THE EFFECT OF OSTEOPATHIC TREATMENT ON CHRONIC NONSPECIFIC NECK PAIN
Acronym: Osteopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Rumeli University (Other)
Responsible Party: Principal Investigator, Ozden Baskan, Assist.Prof, Istanbul Rumeli University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-53938333-050-45260
Record Dates: First submitted 2025-11-21; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Nonspesific Neck Pain
Keywords: Osteopathic Manipulative Treatment; Nonspesific neck pain; Manual Therapy; disability; Physical therapy
MeSH Terms: interventions — Manipulation, Osteopathic

STUDY DESIGN:
Intervention Model Description: This study uses a parallel-group, randomized design in which participants with nonspecific neck pain are assigned to one of two intervention arms. Both groups receive a standard physical therapy protocol, while the experimental group additionally receives a combination of osteopathic techniques, including myofascial release, trigger point therapy, craniosacral osteopathy, visceral osteopathy, osteopathic manipulation, and harmonic mobilization.
  All participants attend four weekly treatment sessions. Outcome assessments are conducted before the first session (baseline) and after the last session (post-intervention). These assessments include pain intensity (VAS), functional status (NDI), quality of life (SF-36), cervical muscle strength, and cervical range of motion. The outcomes assessor is blinded to group allocation to minimize assessment bias.
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor was blinded to group allocation throughout all pre- and post-treatment evaluations. Participants and intervention providers were not blinded due to the nature of the treatments.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Osteopathic treatment and Physical Therapy (Experimental): Receives a combination of osteopathic techniques (myofascial release, trigger point therapy, craniosacral osteopathy, visceral osteopathy, osteopathic manipulation, and harmonic mobilization) in addition to the standard physical therapy protocol (TENS therapy, infrared therapy, and exercise program). Participants received 4 sessions of treatment, once a week.
  Interventions: Procedure: Osteopathic treatment; Procedure: Standard Physical Therapy protocol
- Standard Physical Therapy Protocol (Active Comparator): Participants in this group receive only the standard physical therapy protocol, which includes TENS therapy, infrared therapy, and an exercise program. All participants attend four weekly treatment sessions. Outcome assessments, including pain (VAS), function (NDI), quality of life (SF-36), muscle strength, and cervical range of motion, are conducted before and after the intervention period. The outcomes assessor is blinded to group allocation.
  Interventions: Procedure: Standard Physical Therapy protocol

INTERVENTIONS:
Procedure: Osteopathic treatment — This intervention includes a combination of osteopathic techniques, including myofascial release, trigger point therapy, craniosacral osteopathy, visceral osteopathy, osteopathic manipulation, and harmonic mobilization. Participants receive four weekly sessions, each lasting 45-60 minutes. This intervention is provided in addition to the standard physical therapy protocol.
  Arms: Osteopathic treatment and Physical Therapy
Procedure: Standard Physical Therapy protocol — TENS therapy, infrared therapy, and exercise program.

SUMMARY:
This study evaluates whether adding osteopathic treatment to standard physical therapy improves outcomes in adults with nonspecific neck pain. Forty participants are randomly assigned to two groups: one group receives osteopathic techniques (myofascial release, trigger point therapy, craniosacral osteopathy, visceral osteopathy, osteopathic manipulation, and harmonic mobilization) in addition to standard physical therapy (TENS, infrared, and exercise), while the other group receives only standard physical therapy. All participants attend four weekly sessions. Pain, function, quality of life, muscle strength, and cervical range of motion are assessed before and after treatment. The outcomes assessor is blinded to group allocation. This study aims to determine whether osteopathic interventions provide additional benefits over standard physical therapy.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with nonspecific neck pain for at least three months.
* Pain of musculoskeletal origin.
* Adults aged 18-65 years.
* No analgesic medication taken within the previous 24 hours.

Exclusion Criteria:

* Neck pain due to trauma or injury.
* Presence of osteoporosis or fracture risk.
* Inflammatory or rheumatic diseases.
* Presence of psychological disorders.
* Any systemic disease affecting the musculoskeletal system.
* Use of corticosteroid-containing medications.
* Diagnosis of tumor or cancer.
* Inability to complete the treatment process.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-11-12 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | Baseline and immediately after 4 weekly treatment sessions (4 weeks total)
  Outcome Measure: Pain Intensity Time Frame: Baseline and after 4 weeks (post-intervention) Description: Change in pain level measured using the Visual Analog Scale (VAS) in participants with nonspecific neck pain. The Visual Analog Scale (VAS), a 0-10 scale where 0 indicates no pain and 10 indicates the worst possible pain.

SECONDARY OUTCOMES:
Functional status | Time Frame: Baseline and after 4 weekly treatment sessions (4 weeks total)
  Functional Status Description: Change in functional status measured using the Neck Disability Index (NDI). The NDI consists of 10 items, each scored 0-5, with a total score ranging from 0 (no disability) to 50 (maximum disability). Scores can be converted to a percentage, with higher percentages indicating a greater degree of disability.
Life quality | Baseline and after 4 weekly treatment sessions (4 weeks total)
  Change in health-related quality of life measured using the SF-36 Quality of Life Scale.SF-36 consists of 36 items grouped into 8 domains: physical functioning, role limitations due to physical health, role limitations due to emotional problems, energy/fatigue, emotional well-being, social functioning, pain, and general health. Each domain is scored 0-100, with higher scores indicating better health status or quality of life.
Muscle strength | Baseline and after 4 weekly treatment sessions (4 weeks total)
  Change in cervical and shoulder muscle strength assessed using standardized manual muscle testing. Each muscle group is scored 0-5, where 0 = no contraction and 5 = normal strength against full resistance. Higher scores indicate stronger muscles.
Cervical Range of Motion (ROM) | Baseline and after 4 weekly treatment sessions
  Change in cervical spine range of motion measured using a goniometer. ROM is recorded in degrees for flexion, extension, lateral bending, and rotation. Higher values indicate greater mobility.

CONTACTS AND LOCATIONS:
Locations (1):
- the Fiz-Em Healthy Life Counseling Center, Muğla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) from this study will not be shared because the dataset contains sensitive patient health information, and participants did not provide consent for public data sharing.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-11-12): https://cdn.clinicaltrials.gov/large-docs/22/NCT07260422/Prot_SAP_000.pdf